CLINICAL TRIAL: NCT04225325
Title: Implication for Strategies of Long Term Control of Viral Replication in Patient With Primary HIV Infection (PHI) Treated With Multitarget Antiviral Therapy (MT-ART)
Brief Title: Implication for Strategies of Long Term Control of Viral Replication in Patient With Primary HIV Infection (PHI).
Acronym: P25-INACTION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ADRIANO LAZZARIN, MD (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor-Investigator, ADRIANO LAZZARIN, MD, HEAD OF INFECTIOUS DISEASES CLINIC, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P25-INACTION
Record Dates: First submitted 2019-09-16; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: HIV-1-infection
Keywords: antiretroviral drugs; HIV viral reservoir; HIV acute infection
MeSH Terms: interventions — symtuza

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomised in a ratio 10:10:8 to be treated with one of the three antiretroviral regimens:
  * TDF/FTC 245 mg/200 mg single tablet QD + DRV /cobicistat 800 mg /150 mg single tablet QD (Arm A, standard regimen),
  * TDF/FTC 245 mg/200 mg single tablet QD + DTG 50 mg QD (Arm B, standard regimen).
  * TDF/FTC 245 mg/200 mg single tablet QD + DRV 800 mg /cobicistat single tablet QD + DTG 50 mg QD (Arm C, experimental regimen).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: SYMTUZA (Active Comparator): TAF/FTC 245 mg/200 mg single tablet QD +DRV /cobicistat 800 mg /150 mg single tablet QD
  Interventions: Combination Product: SYMTUZA
- B: DESCOVY+DOLUTEGRAVIR (Active Comparator): TAF/FTC 245 mg/200 mg single tablet QD+DTG 50 mg QD
  Interventions: Combination Product: DESCOVY+DOLUTEGRAVIR
- C: SYMTUZA+DOLUTEGRAVIR (Experimental): TAF/FTC 245 mg/200 mg single tablet QD+DRV/cobicistat single tablet QD + +DTG 50 mg QD
  Interventions: Combination Product: SYMTUZA+DOLUTEGRAVIR

INTERVENTIONS:
Combination Product: SYMTUZA — DESCOVY+REZOLSTA
  Arms: A: SYMTUZA
Combination Product: DESCOVY+DOLUTEGRAVIR — DESCOVY+DOLUTEGRAVIR
  Arms: B: DESCOVY+DOLUTEGRAVIR
Combination Product: SYMTUZA+DOLUTEGRAVIR — DESCOVY+REZOLSTA+DTG
  Arms: C: SYMTUZA+DOLUTEGRAVIR

SUMMARY:
Multicenter, parallel group, randomised, open label, study. Twenty-five clinical centers constituting the InAction network will participate the study.

Eligible patients will be randomised in a ratio 10:10:8 to be treated with one of the three antiretroviral regimens:

* TDF/FTC 245 mg/200 mg single tablet QD + DRV /cobicistat 800 mg /150 mg single tablet QD (Arm A, standard regimen),
* TDF/FTC 245 mg/200 mg single tablet QD + DTG 50 mg QD (Arm B, standard regimen).
* TDF/FTC 245 mg/200 mg single tablet QD + DRV 800 mg /cobicistat single tablet QD + DTG 50 mg QD (Arm C, experimental regimen).

One-hundred-and-twelve PHI subjects will be recruited for this study among those attending the outpatient Clinic of Infectious Diseases, Ospedale San Raffaele and other Italian centres, involved in the INACTION network.

DETAILED DESCRIPTION:
At Screening, potential subjects will perform serology for HIV, ELISA and Western Blot (WB), to assess Fiebig stage:

* Stage I: ELISA negative, WB negative, HIV-1 RNA positive.
* Stage II: ELISA positive for p24, WB negative.
* Stage III: ELISA positive, WB negative.
* Stage IV: ELISA positive, WB undetermined.
* Stage V: ELISA positive, WB partially positive with p31 negative.
* Stage VI: ELISA positive, WB positive, previous HIV negative test within 6 months

On Day 0 (Baseline-BL), within 0-5 days from screening, subjects will:

* perform biochemical and haematological tests, virological test (HIV-1 RNA, tropism test, genotype resistance test), immunological test (CD4+, CD4%, CD8+, CD8%, CD4/CD8).
* Perform anal and nasal brushing
* Perform microbiome
* Have behavioral survey questionnaire administered
* collect an additional sample of blood (80 mL) to perform the following evaluations:

  * HIV-DNA
  * T cells, B cells and DC subsets
  * HLA-A, B and C
  * Inflammatory markers
  * Pharmacokinetic: Ctrough
* start one of the study treatment according to randomization

  * Arm A: TDF/FTC 10 mg/200 mg single tablet QD +DRV /cobicistat 800 mg /150 mg single tablet QD
  * Arm B: TDF/FTC 25 mg/200 mg single tablet QD +DTG 50 mg QD
  * Arm C: TDF/FTC 10 mg/200 mg single tablet QD +DRV/cobicistat single tablet QD +DTG 50 mg QD

In addition, on Day 0 (Baseline-BL), subjects who will sign an additional specific informed consent:

* cerebrospinal fluid (CSF) will be collected to evaluate HIV-1 RNA
* GALT biopsies will be performed in order to allow the evaluation of viral reservoirs.
* Lymph nodes biopsies to evaluate immunological subset Following Day 0, subjects will return for visits at Weeks 2, 4, 8, 12, 24, 36 and 48 or at discontinuation.

HIV-1 RNA levels will be measured and physical examination will be performed at all the scheduled study visits CD4+, CD4%, CD8+, CD8%, CD4/CD8 will be repeated at Weeks 4, 8, 12, 24, 36, 48 or at discontinuation.

Laboratory safety parameters (complete blood count, renal function, hepatic function, lipids and glucidic profile) will be tested at Weeks 4, 8, 12, 24, 36, 48 or at discontinuation.

At week 12 and 48 or at discontinuation, an additional blood sample of 80 mL will be collected to perform the following evaluations:

* HIV-DNA and viral tropism
* T, B and DC cells subsets
* Inflammatory markers At week 2, 4, 8, 12, 24, 36, 48 or at discontinuation a blood sample of 21 mL will be collected for pharmacokinetic of drugs.

At week 12, 48 or discontinuation a stool sample will be collected to evaluate microbioma.

At week 12 and 48 anal brushing and nasal brushing will be performed to evaluate HIVDNA and pharmacokinetic analysis.

At week 12 and 48 behavioral survey questionnaire will be administered to the patient.

At week 12, or at discontinuation, in subjects who will have signed the specific additional informed consent:

* liquor will be collected to evaluate HIV-1 RNA and drugs concentration in central nervous system.
* CSF will be collected to evaluate HIV-1 RNA and drugs concentration in central nervous system.
* GALT biopsies and lymph nodes biopsy will be performed in order to allow the evaluation of viral reservoirs.

Subjects will complete the study when they will reach week 48 on their assigned regimen. At the end of the study, they will continue assigned treatment in arm A and B; if the study will show a superiority of ARM C, the patients in this arm will continue the regimen. In case of non superiority they will be switch to triple therapy. The last patient visit is the last on-study visit or date of death or lost-to follow-up or discontinuation for any reason, whichever occurs last during the conduction of the study.

Considering that the patients' enrollment will last 96 weeks, the overall length of the trial will be 144 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* Subjects must be at least 18 years of age at the time of randomization, of either sex and of any race.
* Primary HIV Infection defined according to Fiebig's classification.
* Subjects must have given written informed consent and must be able to adhere to dose and visit schedules.
* Female subjects of child-bearing potential must agree to use a medically accepted method of contraception.
* Female subjects of child-bearing potential must have a negative serum beta-hCG pregnancy test at Screening, and a negative urine beta-HCG pregnancy test on Day 1 prior to dosing.
* A female, may be eligible to enter and participate in the study if she:

  1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy;
  2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
* Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications;
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 4 for an example listing of approved IUDs);
* Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
* Approved hormonal contraception for subjects randomized to arm B (TDF/FTC + DTG)
* Approved hormonal contraception and a barrier method for subjects randomized to arm A (TDF/FTC +DRV/cobicistat) and C (TDF/FTC +DRV/cobicistat +DTG)
* Any other method with published data showing that the expected failure rate is <1% per year.
* Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of IP. -Approved hormonal contraception for subjects randomized to the treatment groups should be specified.

EXCLUSION CRITERIA:

* Female subjects of childbearing potential who are breastfeeding, pregnant, or planning to become pregnant.
* Subjects with active opportunistic infection or malignancy.
* Subjects positive for Hepatitis B at screening (+HBsAg), or anticipated need for Hepatitis C virus (HCV) therapy during the study.
* Subjects with known liver cirrhosis.
* Subjects with any clinically significant condition or situation other than the condition being studied that, in the opinion of investigator, would interfere with the study evaluations or optimal participation.
* Subjects with allergy/sensitivity to drugs or its excipients.
* History or presence of allergy to the study drugs or their components
* Alanine aminotransferase (ALT) 5 times the upper limit of normal (ULN), OR ALT 3xULN and bilirubin 1.5xULN (with >35% direct bilirubin)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Subject has creatinine clearance of <70 mL/min via Cockroft-Gault method
* Hepatic failure (Child-Plug grade C)
* Use of not modifiable concomitant drugs: carbamazepine, fenitoine, fenobarbital, rifampicine, Hypericum perforatum, dofelitide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-06-14 (Estimated)

PRIMARY OUTCOMES:
the change of total HIV-DNA level from baseline to 48 weeks. | 48 weeks
  The primary objective of the study is to compare the proviral DNA change in patients who started three different antiretroviral treatments.

SECONDARY OUTCOMES:
the proportion of patients with HIV-1 RNA <50 copies/mL | weeks 12, 24 and 48
  proportion of patients with HIV-1 RNA <50 copies/mL at week 24 and week 48;
time to achieve undetectable viral load | week 12 and week 48
  HIV-1 RNA <50 copies/mL
change in HIV-DNA | week 12 and week 48
  the change of total copies/mL OF HIV-DNA level from baseline to 48 weeks
change in HIV-1 RNA in CSF | week 12 and 48
  the change of total copies/mL of HIV-RNA level in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: GIUSEPPE TAMBUSSI, Study Chair — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruzzesi E, Gabrieli A, Bernasconi D, Marchetti G, Calcagno A, Ripamonti D, Antinori A, Squillace N, Cingolani A, Muscatello A, Bandera A, Gori A, Rusconi S, Nozza S; INACTION Study Group. HIV-DNA decrease during treatment in primary HIV-1 infection with three different drug regimens: Italian Network of Acute HIV Infection (INACTION) clinical trial. J Med Virol. 2023 Sep;95(9):e29114. doi: 10.1002/jmv.29114. PMID 37752816